CLINICAL TRIAL: NCT01717729
Title: Hepatocellular Carcinoma Treated With Radiofrequency Ablation With or Without Iodine-125 Implantation: A Prospective Study
Brief Title: Hepatocellular Carcinoma Treated With Iodine-125 Implantation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Second People's Hospital of GuangDong Province (Other)
Responsible Party: Principal Investigator, KaiYun Chen, SURGERY, The Second People's Hospital of GuangDong Province
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ABT-2000-235
Record Dates: First submitted 2012-10-17; First posted 2012-10-30 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: Liver Carcinoma
Keywords: HCC, RFA, Iodine-125, Recurrence
MeSH Terms: conditions — Carcinoma, Hepatocellular; Recurrence | interventions — Radiofrequency Ablation; Iodine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RFA-125I group (Experimental): The combination RFA and 125I (RFA-125I) (n = 68; 42 men, 26 women; mean age, 50.7 years; age range, 29-73 years) In this group, patients were accepted not only radiofrequency ablation (RFA) but also iodine-125.
  Interventions: Procedure: Radiofrequency Ablation; Radiation: iodine
- RFA-only group (Active Comparator): (n = 68; 47 men, 21 women; mean age, 48.9 years; age range, 30-74 years) In tis group,the patient were just peformed radiofrequency ablation alnoe.
  Interventions: Procedure: Radiofrequency Ablation

INTERVENTIONS:
Procedure: Radiofrequency Ablation — For RFA, we used a commercially available system (RF 2000; Radio Therapeutics, Mountain View, Calif) and a needle electrode with a 15-gauge insulated cannula that had 10 hook-shaped expandable electrode tines with a diameter of 3.5 cm at expansion (LeVeen; Radio Therapeutics).The radioactivity per seed ranged from 0.5 to 0.6 millicuries (mCi)
  Other Names: Radio Therapeutics, Mountain View, Calif
Radiation: iodine — The 125I seeds (0.8 mm in diameter and 4.5mm in length) were enclosed in a NiTinol capsule (China Institute of Atomic Energy, Beijing). These seeds could produce 27.4-31.5 keV X-ray and 35.5 Kev γ ray, with a half-life of 59.6 days. The radioactivity per seed ranged from 0.5 to 0.6 millicuries (mCi).
  Other Names: iodine-125 seed
  Arms: RFA-125I group

SUMMARY:
To prospectively evaluate whether use of combined radiofrequency ablation (RFA) and percutaneous iodine-125 (125I) seeds implantation results in better survival compared with use of RFA alone in patients with hepatocellular carcinoma.

DETAILED DESCRIPTION:
This study was local ethical committee approved; all patients gave written informed consent. A total of 136 patients were randomly assigned to undergo RFA-125I (n = 68; 42 men, 26 women; mean age, 50.7 years; age range, 29-73 years) or RFA alone (n = 68; 47 men, 21 women; mean age, 48.9 years; age range, 30-74 years). Patients with viable tumors at computed tomography (CT) 4 weeks after treatment received additional treatment. Rates of local tumor progression and overall survival were evaluated by using Kaplan-Meier and log-rank tests, respectively. The relative prognostic significance of variables in predicting overall survival and the time to tumor recurrence or metastasis were assessed with multivariate Cox proportional hazards regression and logistic regression analyses, respectively.

ELIGIBILITY:
Inclusion Criteria:

(a) age 18-75 years and refusal to undergo surgery; (b) a solitary HCC 7.0 cm in diameter or smaller or multiple (up to three) HCCs 3.0 cm in diameter or smaller; (c) lesions visible at ultrasonography (US), with an acceptable and safe path between the lesion and the skin seen on the US scan; (d) no extrahepatic metastasis; (e) no imaging evidence of tumor invasion into the major portal or hepatic vein branches; (f) no history of encephalopathy, ascites refractory to diuretics, or variceal bleeding; (g) a platelet count of more than 40 000 cells/mm3 and (h) no previous treatment for HCC except liver resection.

Exclusion Criteria:

Exclusion criteria included active thyroid disease, serious concurrent medical illnesses, extrahepatic diseases, previous anticancer treatment before surgery, histologically proved non-HCC tumors and women who were pregnant or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2000-01; Primary Completion 2012-08 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
recurrence rate | up to 6 years
  The primary endpoint was the time to recurrence(TTR) was measured from the date of treatment to the time when the recurrent tumor was first diagnosed. At spiral CT after treatment, residual viable tumor tissue was considered to be present if enhancing areas were seen within the tumor on either arterial phase or portal venous phase images. Depending on the initial random treatment assignment, RFA-125I or RFA alone was repeated. Magnetic resonance (MR) imaging was performed if there was uncertainty at CT as to whether residual viable tumor tissue was present.

SECONDARY OUTCOMES:
One-, 2-, 3-, 4-, and 5-year overall survival rates | up to 6 years
  urvival time was defined as the interval between the first treatment and either death or last follow-up visit.
Complete Ablation | up to 6 years
  At spiral CT 4 weeks after treatment, residual viable tumor tissue was considered to be present if enhancing areas were seen within the tumor on either arterial phase or portal venous phase images.

CONTACTS AND LOCATIONS:
Overall Officials: kai yun chen, phD, Study Chair — The second people's hospital

REFERENCES:
- [Derived] Chen K, Chen G, Wang H, Li H, Xiao J, Duan X, He J, He K, Xiang G. Increased survival in hepatocellular carcinoma with iodine-125 implantation plus radiofrequency ablation: a prospective randomized controlled trial. J Hepatol. 2014 Dec;61(6):1304-11. doi: 10.1016/j.jhep.2014.07.026. Epub 2014 Jul 24. PMID 25064436